CLINICAL TRIAL: NCT06397755
Title: Observational Study of Patients Who Underwent Diagnostic Investigation (Prostate Biopsy) and/or Radical Prostatectomy Surgery.
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Professor, IRCCS San Raffaele
Other Study IDs: 2014-Prostata
Record Dates: First submitted 2023-10-13; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent prostate biopsy and/or radical prostatectomy surgery.
  Interventions: Procedure: Prostate Biopsy and/or Radical Prostatectomy

INTERVENTIONS:
Procedure: Prostate Biopsy and/or Radical Prostatectomy — Prostate Biopsy: procedure to remove samples of suspicious tissue from the prostate Radical Prostatectomy: surgery to remove the prostate gland and seminal vesicles (and sometimes nearby lymph nodes) after a prostate cancer diagnosis

SUMMARY:
This is a single-center, observational, prospective and retrospective study on quality of life and disease status of patients who underwent prostate biopsy and/or radical prostatectomy.

DETAILED DESCRIPTION:
A database was created with the intention of collecting data related to patients who underwent prostate biopsy and/or radical prostatectomy.

Only anamnesis and biopsy procedure data are collected for patients underwent prostate biopsy.

Anamnesis, surgery, histological report and hospitalization data are collected for patients who underwent radical prostatectomy.

Each patient will be followed for 50 years from the date of radical prostatectomy surgery.

Each patient will receive a questionnaire before radical prostatectomy. A follow up questionnaire will be collected after surgery relating to quality of life. The data for each patient will then be transferred to the database itself. The data collected will be handled following the most strict GCPs and privacy norms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suspicious prostate disease who underwent prostate biopsy and/or radical prostatectomy;
* Adult patients > 18 years
* Ability to read and sign the informed consent

Exclusion Criteria:

* Patients < 18 years
* mental or physical disability that may prevent the patient from satisfying the requirements of the protocol
* Inability to read and sign the informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the urology department who need undergo prostate biopsy and/or radical prostatectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2015-01-08 (Actual); Primary Completion 2065-01-08 (Estimated); Study Completion 2065-01-08 (Estimated)

PRIMARY OUTCOMES:
Clinically significant Prostate Cancer | 1 month
  Diagnosis of clinically significant PCa at prostate biopsy
Overall survival | every 6 month after surgery up to 50 years after surgery
  Death by any cause
Cancer-specific mortality | every 6 month after surgery up to 50 years after surgery
  Death from prostate cancer
Biochemical recurrence | every 6 month after surgery up to 50 years after surgery
  PSA >= 0.2 ng/ml in 2 consecutive measures

SECONDARY OUTCOMES:
Erectile function | every 6 month after surgery up to 50 years after surgery
  IIEF-EF >=21
Urinary continence | every 6 month after surgery up to 50 years after surgery
  No pads over a 24 hour period

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No